CLINICAL TRIAL: NCT02915965
Title: A Phase II Trial of Neoadjuvant Chemotherapy for Stage II, III Esophageal Squamous Cell Carcinoma
Brief Title: A Trial of Neoadjuvant Chemotherapy for Stage II, III Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, MD, PHD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESCC01-SUMS6
Record Dates: First submitted 2016-09-23; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Stage II and III Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Surgical Procedures, Operative

ARMS (1):
- DCX and surgery (Experimental): docetaxol 60mg/m2 iv d1 and cisplatin 30mg/m2 iv d1-2 and capecitabine 850mg/m2 bid po d1-14 repeated every 21 days for 4-6 cycles, followed by surgery of Ivor Lewis Esophagectomy
  Interventions: Drug: DCX; Procedure: surgery

INTERVENTIONS:
Drug: DCX — docetaxel, cisplatin and capecitabine
Procedure: surgery — Ivor Lewis Esophagectomy

SUMMARY:
The purpose of this study is to determine whether docetaxel, cisplatin, and capecitabine (DCX) are effective as the neoadjuvant chemotherapy before esophagectomy in patients with loco-regional esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of squamous cell thoracic esophageal carcinoma of Stage II or III, which is potentially resectable.
2. Patients must not have received any prior anticancer therapy.
3. More than 6 months of expected survival.
4. Age ranges from 18 to 70 years.
5. Absolute white blood cells count ≥4.0×109/L, neutrophil ≥1.5×109/L, platelets ≥100.0×109/L, hemoglobin ≥90g/L, and normal functions of liver and kidney.
6. Karnofsky performance status (KPS) of 90 or more.
7. Signed informed consent document on file.

Exclusion Criteria:

1. Patients are diagnosed or suspected to be allergic to docetaxol or cisplatin or capecitabine.
2. Patients with concomitant hemorrhagic disease.
3. Pregnant or breast feeding.
4. Inability to use gastric conduit after esophagectomy because of a prior surgery.
5. Patients with concomitant peripheral neuropathy, whose common toxicity criterion (CTC) status is 2 or even more.
6. Have a prior malignancy other than esophageal carcinoma, carcinoma in situ of the cervix, nonmelanoma skin cancer or cured early stage of prostate cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
overall survival rate | 2 years

SECONDARY OUTCOMES:
Pathologic response rate | 2 years
  Pathologic response rate is defined as tumor regression score
Disease-free survival | 2 years
Incidence of adverse event based on CTCAE 4.0 | 2 years
  Incidence of adverse event in patients during treatment period graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, MD PHD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China